CLINICAL TRIAL: NCT01763047
Title: Evaluation of the Performance of Investigational Contact Lenses in a Presbyopic Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR-5357
Record Dates: First submitted 2012-12-17; First posted 2013-01-08 (Estimated); Results first posted 2016-06-10 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-05

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- etafilcon A/lotrafilcon B (Active Comparator): Subjects were randomized to one of two lens wear sequences. Subject randomized to this sequence first wore the etafilcon A lens and then wore the lotrafilcon B lens.
  Interventions: Device: etafilcon A; Device: lotrafilcon B
- lotrafilcon B/etafilcon A (Active Comparator): Subjects were randomized to one of two lens wear sequences. Subject randomized to this sequence first wore the lotrafilcon B lens and then wore the etafilcon A lens.
  Interventions: Device: etafilcon A; Device: lotrafilcon B

INTERVENTIONS:
Device: etafilcon A — To be worn in a daily wear modality for a minimum of 6 hours per day.
Device: lotrafilcon B — Lenses will be worn in a reuseable modality; cleaned and disinfected each night.
  Other Names: AirOptix Aqua Multifocal

SUMMARY:
The objective of this study is to evaluate the performance of a novel multifocal lens system.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Subjects must appear able and willing to adhere to the instructions set forth in the clinical protocol.
3. Subjects must be between 40 and 70 years of age.
4. Subjects' spherical equivalent distance refraction must be in the range of -3.75 to +3.75 in each eye.
5. Subjects' refractive cylinder must be less than or equal to 0.75D in each eye.
6. Subjects' ADD power must be in the range of +0.75 to +2.50D in each eye.
7. Subjects' must have the best corrected visual acuity of 20/20-3 or better in each eye.
8. Subjects' should own a wearable pair of spectacles.
9. Subjects' must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month or more duration).
10. Subjects' must respond positively to at least on symptom on the "Presbyopis Symptoms Questionnaire" or already be wearing a presbyopic contact lens correction (e.g. reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.).

Exclusion Criteria:

1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
2. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
3. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear.
4. Any previous intraocular surgery (e.g. radial keratotomy, PRK, LASIK, etc.)
5. Any grade 3 or greater slit lamp findings (e.g. edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) which may contraindicate contact lens wear.
6. Any ocular infection.
7. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
8. History of binocular vision abnormality or strabismus.
9. Any infectious disease (e.g. hepatitis, tuberculosis) or contagious immunosuppressive disease (e.g. HIV).
10. History of diabetes.
11. Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Mission Viejo, California
  - RPS, Jacksonville, Florida
  - Jacksonville, Florida
  - Saint Augustine, Florida
  - Tallahassee, Florida
  - Winter Park, Florida
  - Roswell, Georgia
  - Lutherville, Maryland
  - Closter, New Jersey
  - New York, New York
  - Denver, North Carolina
  - Athens, Ohio
  - Kingston, Pennsylvania
  - Warwick, Rhode Island
  - Memphis, Tennessee
  - Amarillo, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - Salem, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study enrolled a total of 298 subjects. Subjects were stratified as either Hyperopes or Myopes, which was determined by their sphere power. Of the enrolled subjects 22 did not meet the eligibility criteria and 276 subjects were randomized a study lens. Of the randomized subjects 29 were discontinued and 247 subjects completed the study.
Groups:
- Etafilcon A/ Lotrafilcon B: Subjects were randomly assigned to one of two possible lens sequences. Subjects first received the etafilcon A lens and then received the lotrafilcon B lens.
- Lotrafilcon B/ Etafilcon A: Subjects were randomly assigned to one of two possible lens sequences. Subjects first received the lotrafilcon B lens and then received the etafilcon A lens.
Period: Period 1
Arm/Group | Etafilcon A/ Lotrafilcon B | Lotrafilcon B/ Etafilcon A
Started | 139 | 137
Myopes | 77 | 76
Hyperopes | 62 | 61
Completed | 130 | 126
Not Completed | 9 | 11
Not completed — Test Article Not Available | 4 | 1
Not completed — Protocol Violation | 4 | 4
Not completed — No Longer Meets Eligibility criteria | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Unsatisfactory Visual Response | 0 | 3
Not completed — Lens Power Not Available | 0 | 1
Not completed — Study Site office Closed | 0 | 1
Period: Period 2
Arm/Group | Etafilcon A/ Lotrafilcon B | Lotrafilcon B/ Etafilcon A
Started | 130 | 126
Myopes | 74 | 72
Hyperopes | 56 | 54
Completed | 126 | 121
Not Completed | 4 | 5
Not completed — Lens Discomfort | 1 | 0
Not completed — No longer meets Eligibility Criteria | 1 | 0
Not completed — Study Site office Closed | 1 | 1
Not completed — Unsatisfactory Visual Response | 1 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Unsatisfactory lens Fitting | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized subjects that were dispensed at least one study lens.
Groups:
- Etafilcon A/ Lotrafilcon B: Subjects were randomly assigned to one of two possible lens sequences. Subjects first received the etafilcon A and then received the lotrafilcon B.
- Lotrafilcon B/ Etafilcon A: Subjects were randomly assigned to one of two possible lens sequences. Subjects first received the lotrafilcon B and then received the etafilcon A.
- Total: Total of all reporting groups
Arm/Group | Etafilcon A/ Lotrafilcon B | Lotrafilcon B/ Etafilcon A | Total
Number analyzed (Participants) | 139 | 137 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.49 (6.626) | 50.90 (6.775) | 50.69 (6.691)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 108 | 216
  Male | 31 | 29 | 60
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 2 | 3 | 5
  Black or African American | 13 | 10 | 23
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  White | 121 | 123 | 244
  other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 139 | 137 | 276

OUTCOME MEASURES:

1. Primary Outcome: Binocular Distance Visual Acuity (LogMAR)
Description: Distance time controlled LogMAR Visual Acuity was carried out binocularly with high luminance and high contrast, at 4m under 250 cd/m^2. The test was presented under the condition High luminance (250 cd/m^2) High Contrast (90%)
Time Frame: 8-12 days post wear
Population: The analysis population consists of subjects that completed all study visits without a major protocol deviation. The analysis was conducted on each lens and strata.
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Etafilcon A: Subjects that were dispensed the etafilcon A lens during either the first or second period of the study.
- Lotrafilcon B: Subjects that were dispensed the lotrafilcon B lens during either the first or second period of the study.
Arm/Group | Etafilcon A | Lotrafilcon B
Number analyzed (Participants) | 207 | 207
LogMAR
  Hyperopes, N=91, 91 | -0.068 (0.0885) | -0.058 (0.0867)
  Myopes, N=116, N=116 | -0.109 (0.0826) | -0.107 (0.0835)

2. Primary Outcome: Binocular Near Visual Acuity (logMAR)
Description: Near time controlled LogMAR Visual Acuity was carried out binocularly using High lumiance and High Contrast, at 40cm under 250 cd/m^2. The test was presented under the condition High Luminance (250cd/m^2) High Contrast (90%).
Time Frame: 8-12 days post wear
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Lotrafilcon B: Subjects that were dispensed the lotrafilcon B during either the first or second period of the study.
Arm/Group | Etafilcon A | Lotrafilcon B
Number analyzed (Participants) | 207 | 207
LogMAR
  Hyperopes, N=91, N=91 | 0.063 (0.1070) | 0.082 (0.1316)
  Myopes, N=116, N=116 | 0.048 (0.1106) | 0.043 (0.0975)

3. Primary Outcome: Percentage of Eyes With Corneal Staining Grade 3 or Higher
Description: Corneal staining was evaluated in 5 corneal regions (Central, Inferior, Nasal, Temporal and Superior) using Sodium Fluorescein strips. The Fluorescien strip was lightly placed on the subject's inferior palpebral conjunctiva. The corneal Staining was graded using the scale Grade 0: No Staining, Grade 1: Trace(Minimal superficial staining or stippling), Grade 2: Mild (Regional or diffuse punctate staining), Grade 3:Moderate(Significant dense coalesced staining, corneal abrasion or foreign body tracks.), Grade 4 Severe(Severe abrasions greater than 2 mm in diameter, ulcerations, epithelial loss, or full thickness abrasion.). The data was dichotomized into two group subjects with grade 3 or higher and those subjects with less than Grade 3 for the maximum grade of corneal staining across all 5 regions.
Time Frame: 8-12 days post wear
Population: The analysis population consists of subjects that completed all study visits without a major protocol deviation.The analysis was conducted on subject eyes for each lens and strata.
Measure: Number; unit: Percentage of Subject Eyes
Units Other Than Participants: Subject Eyes
Groups:
- Etafilcon A: Subjects that were dispensed the etafilcon A during either the first or second period of the study. Subjects were then stratified by sphere power as either Hyperopes or Myopes.
- Lotrafilcon B: Subjects that were dispensed the lotrafilcon B during either the first or second period of the study. Subjects were then stratified by sphere power as either Hyperopes or Myopes.
Arm/Group | Etafilcon A | Lotrafilcon B
Number analyzed (Participants) | 207 | 207
Number analyzed (Subject Eyes) | 414 | 414
Percentage of Subject Eyes
  Hyperopes, N=182, N=182 | 0.0 | 0.0
  Myopes, N=232, N=232 | 0.0 | 0.0

4. Primary Outcome: Percentage of Eyes With Limbal Conjunctival Redness Grade 3 or Higher
Description: The Limbus refers to the 1 to 2mm wide zone of conjunctiva and underlying tissue adjacent to where the cornea joins the sclera. Limbal Conjuctival Redness was graded in 4 regions (Nasal, Temporal, Inferior and Superior) using the Efron Grading Scale in 1 unit increments. Grade 0: Normal, Grade 1: Trace, Grade 2: Mild, Grade 3: Moderate, Grade 4: Severe. The data was dichotomized into two group subjects with grade 3 or higher Limbal Conjuctival Redness, and those subjects with less than Grade 3 for the maximum grade of all 4 regions.
Time Frame: 8-12 days post wear
Population: The Analysis population consists of subjects that completed all study visits without a major protocol deviation. The analysis was conducted on subject eyes for each lens and strata.
Measure: Number; unit: Percentage of Subject Eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Etafilcon A | Lotrafilcon B
Number analyzed (Participants) | 207 | 207
Number analyzed (Subject Eyes) | 414 | 414
Percentage of Subject Eyes
  Hyperopes, N=182, N=182 | 0.0 | 0.0
  Myopes, N=232, N=232 | 0.0 | 0.0

5. Primary Outcome: Percentage of Eyes With Bulbar Conjunctival Redness Grade 3 or Higher
Description: Bulbar Conjunctival Injection was assessed in 4 regions (Nasal, Temporal, Inferior and Superior) using an Efron Grading scale by 1 unit increments. Grade 0: Normal, Grade 1: Trace, Grade 2: Mild, Grade 3: Moderate, Grade 4:Severe. The data was dichotomized into two group subjects with grade 3 or higher Conjunctival injection, and those subjects with less than Grade 3 for the maximum grade of all 4 regions.
Time Frame: 8-12 days post wear
Population: as for outcome 4
Measure: Number; unit: Percentage of Subject Eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Etafilcon A | Lotrafilcon B
Number analyzed (Participants) | 207 | 207
Number analyzed (Subject Eyes) | 414 | 414
Percentage of Subject Eyes
  Hyperopes, N=182, N=182 | 0.0 | 0.0
  Myopes, N=232, N=232 | 0.0 | 0.0

6. Primary Outcome: CLUE Overall Quality of Vision Using the Contact Lens User Experience (CLUE)TM Questionnaire
Description: CLUE Overall Quality of Vision is assessed using the Contact Lens User Experience (CLUE)TM questionnaire. CLUE is a validated patient-reported outcomes questionnaire to assess patient experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. 97% of the scores fall within 0 and 120 (mean +/-3XSD).
Time Frame: 8-12 days post wear
Population: The analysis consists of subjects that completed all study visits without a major protocol deviation. The analysis was conducted on each lens and strata.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etafilcon A | Lotrafilcon B
Number analyzed (Participants) | 207 | 207
units on a scale
  Hyperopes, N=91, N=91 | 46.48 (18.834) | 44.79 (18.439)
  Myopes, N=116, N=116 | 47.74 (19.279) | 50.17 (20.433)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study- approximately 3 months
Groups:
- Test (Etafilcon A): Subjects that were dispensed the Test lens (etafilcon A) during either the first or second period of the study.
- Control (Lotrafilcon B): Subjects that were dispensed the Control lens (lotrafilcon B) during either the first or second period of the study.
Arm/Group | Test (Etafilcon A) | Control (Lotrafilcon B)
Serious Adverse Events (participants affected / at risk) | 0/276 | 0/276
Other Adverse Events (participants affected / at risk) | 0/276 | 0/276

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days